CLINICAL TRIAL: NCT04149496
Title: A Prospective Series of IVF Cases Utilizing in Vitro Maturation (IVM) With Low Cost Priming, Enhanced Oocyte Recovery, and Delayed Embryo Transfer Using a Subsequent Frozen Embryo Transfer Cycle
Brief Title: IVM With Low Cost Priming, Enhanced Oocyte Recovery, and Delayed Transfer
Acronym: IVMprt
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bruce Rose, MD (Other)
Responsible Party: Sponsor-Investigator, Bruce Rose, MD, principal investigator, Brown Fertility
Organization: Brown Fertility (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-49
Record Dates: First submitted 2019-07-09; First posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Polycystic Ovary Syndrome
Keywords: IVM; in vitro maturation; polycystic ovarian syndrome; PCOS; Steiner-Tan needle; oocyte maturation
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — In Vitro Oocyte Maturation Techniques

STUDY DESIGN:
Intervention Model Description: Prospective series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- All (Experimental): Patients requiring IVF treatment with PCOS or a PCO pattern in their ovaries who wish to undertake IVM (as a variant of their IVF procedure)
  Interventions: Combination Product: in vitro maturation of oocytes

INTERVENTIONS:
Combination Product: in vitro maturation of oocytes — Immature oocytes (rather than mature oocytes) are harvested as in IVF. These oocytes are allowed to mature in the laboratory before fertilization

SUMMARY:
A protocol was developed to improve pregnancy results after IVM compared to results from studies in the literature. Differences from most published protocols include the use of the Steiner-Tan needle to optimize oocyte environment during oocyte retrieval, use of oral medications and very low doses of FSH, and delayed embryo transfer during subsequent warmed cryo-preserved embryo transfer. Eligible patient have a PCO pattern in their ovaries during transvaginal ultrasound.

DETAILED DESCRIPTION:
All participants are candidates for IVF having PCOS or having PCO patterns in their ovaries who wish to undertake IVM for the potential advantages that it holds. All cycles are proceeded by oral contraceptive use for cycle scheduling purposes. Priming is done with oral letrozole with the addition of 25-75 IU daily starting after 2 days of letrozole. HCG is given when several follicle have diameters 8 mm or greater and no follicles have diameters greater than 13 mm. Oocyte retrieval is done approximately 38 hours later. A Steiner-Tan needle is used for oocyte retrieval in a manner that minimizes the amount of time that an oocyte is out of the ovary and not in a controlled laboratory environment. Oocytes are assessed for maturity for up to 48 hours post retrieval. If mature, oocytes are injected with sperm using ICSI. Embryos are grown to blastocysts and all blastocyst are vitrified. Warmed cryo-preserved blastocyst are transferred using routine IVF protocols during a subsequent cycle.

ELIGIBILITY:
Inclusion Criteria:

* PCO pattern with > 25 antral follicles
* AMH > 3.5

Exclusion Criteria:

* BMI > 35
* body morphology making transvaginal retrieval difficult or impossible
* complicating medical condition making pregnancy or IVF relatively contra-indicated

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — genetic female with ovaries and uterus
Enrollment: 300 (Estimated)
Dates: Start 2019-05-10 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of treated patients having a clinical pregnancy | 12 weeks post transfer
  ultrasound evidence of pregnancy in uterus or tissue evidence of pregnancy
Percentage of treated patients having an ongoing pregnancy | 10 months post transfer
  pregnancy with cardiac activity (by history or observations) after 12 weeks

SECONDARY OUTCOMES:
Percentage of retrieved oocytes which matured per patient | 2 days post retrieval
  proportion of retrieved oocytes which are mature (polar body present) within 48 hours of retrieval
Percentage of retrieved oocytes which fertilized per patient | 4 days post retrieval
  proportion of mature oocytes which display pronuclei
Percentage of fertilized oocytes which divided | 6 days post retrieval
  proportion of fertilized oocytes which become 2 or more cells
Percentage of fertilized oocytes which became blastocysts per patient | 8 days post retrieval
  proportion of fertilized oocytes which form a fluid filled cavity
Percentage of patients who have a biochemical pregnancy after therir first transfer | 28 days post transfer
  proportion of patients with an hCG level greater than 5 measured post first transfer

OTHER OUTCOMES:
Number of clinical pregnancies from subsequent transfers | up to one year after transfer of last patient enrolled
  Number of clinical pregnancies from all blastocyst transfers related to the retrieval
Number of ongoing pregnancies from subsequent transfers | up to one year after transfer of last patient enrolled
  Number of ongoing pregnancies from blastocyst transfers related to the retrieval

CONTACTS AND LOCATIONS:
Overall Officials: Bruce I Rose, MD, PhD, Principal Investigator — Brown Fertility
Locations (1):
- Brown Fertility, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rose BI. The potential of letrozole use for priming in vitro maturation cycles. Facts Views Vis Obgyn. 2014;6(3):150-5. PMID 25374658
- [Background] Rose BI: The case for more active management of endometrial development in IVM: Decreasing the miscarriage rate and increasing the clinical pregnancy rate. Journal of Reproductive Endocrinology and Infertility, 14: 1-6, 2016
- [Background] Rose BI, Laky D. A comparison of the Cook single lumen immature ovum IVM needle to the Steiner-Tan pseudo double lumen flushing needle for oocyte retrieval for IVM. J Assist Reprod Genet. 2013 Jun;30(6):855-60. doi: 10.1007/s10815-013-0006-1. Epub 2013 May 5. PMID 23644950